CLINICAL TRIAL: NCT06728306
Title: Acute Impact of Virtual Reality-Based Relaxation and Exergaming Compared to Traditional Relaxation on Primary Dysmenorrhea Symptoms: A Randomised Controlled Trial
Brief Title: Virtual Reality-Based Relaxation and Exergaming vs. Traditional Relaxation for Primer Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Muhammed Şeref Yıldırım, Principle Investigator, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TU-FTR-MŞY-002; 1919B012219298 (Other Grant/Funding Number: The Scientific and Technological Research Council of Turkey)
Record Dates: First submitted 2024-12-05; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Primary Dysmenorrhea
Keywords: Exercise Therapy; Pain Management; Primary Dysmenorrhea; Progressive Muscle Relaxation; Virtual Reality
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immersive Virtual Reality Based Relaxation (Experimental)
  Interventions: Behavioral: Immersive Virtual Reality-Based Relaxation
- Non-Immersive Virtual Reality Based Exergaming (Experimental)
  Interventions: Behavioral: Non-immersive VR-Based Exergaming
- Traditional Jacobson's Relaxation (Active Comparator)
  Interventions: Behavioral: Jacobson's Relaxation

INTERVENTIONS:
Behavioral: Immersive Virtual Reality-Based Relaxation — Participants experienced a 20-minute immersive relaxation session using the virtual reality headset and the "Nature Treks" application, while seated comfortably. Participants were instructed to select the natural environment they found most relaxing from options such as "Blue Ocean," "Orange Sunset," "Violet Down," "White Winter," and "Green Meadows," and spent 20 minutes immersed in their chosen virtual environment.
  Arms: Immersive Virtual Reality Based Relaxation
Behavioral: Non-immersive VR-Based Exergaming — Participants engaged in a 20-minute calisthenic exercise session guided by the Kinect Adventures game on the Xbox Kinect 360 system. The exercise session consisted of playing two rounds each of the game segments "20,000 Leaks", "Reflex Ridge", and "River Rush", each lasting approximately 3 minutes
  Arms: Non-Immersive Virtual Reality Based Exergaming
Behavioral: Jacobson's Relaxation — Participants underwent 20 minutes of progressive relaxation training as developed by Dr. Jacobson. The training involves a series of deep diaphragmatic breaths followed by the systematic tensing and relaxing of 16 major muscle groups throughout the body. Participants were guided through the exercise by an approximately 20-minute audio recording prepared by a psychologist and available online
  Arms: Traditional Jacobson's Relaxation

SUMMARY:
The goal of this clinical trial is to investigate the acute effects of virtual reality-based relaxation (immersive VR relaxation) and exergaming (non-immersive VR) compared to traditional Jacobson's relaxation on symptoms of primary dysmenorrhea (PD) in women aged 18-30 years with regular menstrual cycles. The main questions it aims to answer are:

Does immersive VR relaxation reduce abdomino-pelvic pain and menstrual symptom severity more effectively than Jacobson's relaxation? Does non-immersive VR exergaming provide better pain relief and symptom management compared to traditional relaxation methods?

Hypotheses:

Immersive VR relaxation will result in significantly greater reductions in abdomino-pelvic pain and menstrual symptom severity compared to traditional relaxation.

Non-immersive VR exergaming will also provide better outcomes in pain and symptom management compared to traditional relaxation.

Researchers will compare immersive VR relaxation, non-immersive VR exergaming, and Jacobson's relaxation (control group) to determine the relative effectiveness of each intervention.

Participants will:

Engage in a 20-minute session of one of the assigned interventions. Complete questionnaires on abdomino-pelvic pain, menstrual symptoms, and perceived effectiveness.

Participate in follow-up assessments for sleep quality during menstruation. This study aims to explore innovative, technology-driven approaches for managing menstrual symptoms and their effectiveness relative to traditional methods.

DETAILED DESCRIPTION:
This study seeks to address this gap by investigating whether these innovative approaches can provide superior symptom relief. By evaluating pain intensity, symptom severity, and perceived effectiveness, this research will provide valuable insights into the feasibility and advantages of integrating technology into dysmenorrhea management.

ELIGIBILITY:
Inclusion Criteria:

* women aged 18-30 with no pregnancy history.
* a regular menstrual cycle (28 ± 7 days) over the past 6 months
* menstrual pain with a Visual Analog Scale score >4 during this period

Exclusion Criteria:

* regular medication use or medical treatment during the study (e.g., oral contraceptives, antidepressants).
* recent musculoskeletal trauma or surgery.
* intrauterine device use or pathological conditions/ultrasound findings of secondary dysmenorrhea
* consumption of painkillers, alcohol, recreational drugs, or similar substances within the last 48 hours.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-02-04 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Abdomino-Pelvic Pain İntensity (APPI) | Immediately before and immediately after the 20-minute intervention session
  Visuel Analogue Scale was used to measure abdomino-pelvic pain intensity. A 10 cm line was labeled with "0 cm" indicating no pain and "10 cm" representing unbearable pain at each end. Participants were asked to indicate their pain level by either drawing a line, placing a dot, or marking a point along the scale. Pain assessments were made for the most painful menstrual day and abdomino-pelvic pain on the intervention day.
Menstruation-Related Symptoms | Immediately before and immediately after the 20-minute intervention session
  The Daily Symptom Rating Scale (DSRS), a 17-item self-report tool, was used to assess the intensity of various menstrual symptoms, including pain, mood swings, and physical discomfort. Each symptom was rated on a scale from 0 (no symptoms) to 5 (severe), with higher scores indicating greater symptom severity. The Turkish version of the scale has been validated and shown to be reliable .

SECONDARY OUTCOMES:
Sleep Quality | The morning following the intervention and the morning of the most painful day during the subsequent menstrual cycle.
  Richard Campbell Sleep Questionairre was used to assess sleep quality on the night following the intervention and during a non-intervention menstruation day. The six-item self-report questionnaire, validated in Turkish, evaluates aspects such as sleep depth, latency, frequency of awakenings, and overall quality, with higher scores indicating better sleep quality.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Trakya University, Edirne, İskender
  - Trakya University, Edirne

IPD SHARING:
Plan to Share IPD: No